CLINICAL TRIAL: NCT05217251
Title: The Values of Electroencephalography (EEG) Alterations of Uterine Contractions in the First Stage of Labor Predicting Postpartum Depression: a Prospective Cohort Study
Brief Title: EEG Alterations of Uterine Contractions in the First Stage of Labor Predicting Postpartum Depression
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Maternal EEG monitoring
Record Dates: First submitted 2022-01-16; First posted 2022-02-01 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-01

CONDITIONS: Postpartum Depression
Keywords: electroencephalogram; uterine contractions; in the first stage of labor; Postpartum Depression; frontal alpha asymmetry
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- exposed group: Parturient women will be identified with frontal alpha asymmetry based on EEG monitoring of uterine contractions in the first stage of labor and will then be allocated to vaginal delivery with alpha asymmetry group in hospital.
  Interventions: Other: frontal alpha asymmetry in EEG
- control group: Parturient women will be identified without frontal alpha asymmetry based on EEG monitoring of uterine contractions in the first stage of labor and will then be allocated to vaginal delivery without alpha asymmetry group in hospital.
  Interventions: Other: frontal alpha asymmetry in EEG

INTERVENTIONS:
Other: frontal alpha asymmetry in EEG — frontal alpha asymmetry based on EEG monitoring of uterine contractions in the first stage of labor. The power spectra will be log-transformed and averaged across the frontal left (FL) channels (FP1, F3, F7) and frontal right (FR) channels (FP2, F4, F8). A higher power spectrum value indicates lower neural activity. Frontal asymmetry (FA) power scores are calculated as follows, FA = (FR-FL)/(FR+FL). A positive FA value shows greater neural activity in the left frontal lobe than right frontal neural activity (relative left frontal asymmetry), while its negative value shows oppositely.

SUMMARY:
Severe uterine contractions in labor can trigger emotional disorders including postpartum depression in women during the puerperium. Numerous studies have shown that resting frontal electroencephalogram (EEG) asymmetry is closely related to depression. Therefore, the investigators hypothesize that the frontal alpha asymmetry in EEG during uterine contractions in the first stage of labor be associated with the risk level of postpartum depression. The objective of this research is to investigate, in a 1-year period, the incidence of postpartum depression in natural birth mothers in relation to frontal alpha asymmetry in EEG during uterine contractions and resting state.

DETAILED DESCRIPTION:
Severe uterine contractions in labor can trigger emotional disorders including postpartum depression in women during the puerperium. It is characterized by lack of motivation and behavioral changes, potentially producing serious negative consequences for offspring.

In addition, EEG alpha asymmetry is one of the commonly studied biomarkers for depression. There are multiple previous studies regarding the symmetry of EEG in left and right brain hemispheres, especially at frontal electrodes. Besides, there are many other EEG indicators that predict depression which are also likely to be strong contributors to postpartum depression.

The objective of study is to investigate if there is any association between EEG alterations of uterine contractions in the first stage of labor and factors that are associated with postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* parturient women with a singleton pregnancy;
* capable of understanding the research requirements and willing to cooperate with the study instructions;
* aged 18-45;
* American Society of Anesthesiologists(ASA) physical status I or II;
* right handed;
* not taking any drug known to influence the EEG;
* EPDS scale (Edinburgh Postnatal Depression Scale, EPDS) is used in the last prenatal examination in outpatient clinics , with scores < 10;
* informed consent is gained from all individual subjects taking part in the study.

Exclusion Criteria:

* history of neurological or psychiatric disease;
* personality disorder;
* cerebral disease;
* epidural anesthesia contraindication;
* multiparous pregnancy.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will consist of parturient women who plan a vaginal delivery in Zhujiang hospital .
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of depression in 12 months after childbirth. | up to 12 months after childbirth.
  Postpartum depression in 12 months is diagnosed by using Edinburgh Postpartum Depression Scale (EPDS) by a research assistant. the threshold of postpartum depression is defined as a score of ≥10.The EPDS is a 10-item self-report scale to screen for Postnatal Depression. The EPDS is found to have satisfactory sensitivity and specificity, and is also sensitive to change in the severity of depression over time. Each question is on a scale of 0 to 3. The EPDS has a score range between 0 to 30, with a higher score reflecting higher symptom severity in depression.

SECONDARY OUTCOMES:
The score of pain in 12 months after childbirth | up to 12 months after childbirth.
  The score of pain at in 12 months after childbirth is assessed by using a Visual Analogue Scale (an 10-point scale where 0 indicates no pain and 10 the worst pain).The Visual Analogue Scale is a self-reported scale consisting of a horizontal or vertical line, usually 10 centimeters long (100 mm) anchored at the extremes by two verbal descriptors referring to the pain status . An introductory question asks the patient to express that best refers to her pain.

CONTACTS AND LOCATIONS:
Overall Officials: HongFei Zhang, MD PhD, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howard LM, Molyneaux E, Dennis CL, Rochat T, Stein A, Milgrom J. Non-psychotic mental disorders in the perinatal period. Lancet. 2014 Nov 15;384(9956):1775-88. doi: 10.1016/S0140-6736(14)61276-9. Epub 2014 Nov 14. PMID 25455248
- [Background] O'Hara MW, McCabe JE. Postpartum depression: current status and future directions. Annu Rev Clin Psychol. 2013;9:379-407. doi: 10.1146/annurev-clinpsy-050212-185612. Epub 2013 Feb 1. PMID 23394227
- [Background] Deng CM, Ding T, Li S, Lei B, Xu MJ, Wang L, Xu SC, Yang HX, Sun XY, Li XY, Ma D, Wang DX. Neuraxial labor analgesia is associated with a reduced risk of postpartum depression: A multicenter prospective cohort study with propensity score matching. J Affect Disord. 2021 Feb 15;281:342-350. doi: 10.1016/j.jad.2020.12.027. Epub 2020 Dec 8. PMID 33348177
- [Background] Tian T, Li Y, Xie D, Shen Y, Ren J, Wu W, Guan C, Zhang Z, Zhang D, Gao C, Zhang X, Wu J, Deng H, Wang G, Zhang Y, Shao Y, Rong H, Gan Z, Sun Y, Hu B, Pan J, Li Y, Sun S, Song L, Fan X, Li Y, Zhao X, Yang B, Lv L, Chen Y, Wang X, Ning Y, Shi S, Chen Y, Kendler KS, Flint J, Tian H. Clinical features and risk factors for post-partum depression in a large cohort of Chinese women with recurrent major depressive disorder. J Affect Disord. 2012 Feb;136(3):983-7. doi: 10.1016/j.jad.2011.06.047. Epub 2011 Aug 7. PMID 21824665
- [Background] Purdon PL, Sampson A, Pavone KJ, Brown EN. Clinical Electroencephalography for Anesthesiologists: Part I: Background and Basic Signatures. Anesthesiology. 2015 Oct;123(4):937-60. doi: 10.1097/ALN.0000000000000841. PMID 26275092
- [Background] Koller-Schlaud K, Strohle A, Barwolf E, Behr J, Rentzsch J. EEG Frontal Asymmetry and Theta Power in Unipolar and Bipolar Depression. J Affect Disord. 2020 Nov 1;276:501-510. doi: 10.1016/j.jad.2020.07.011. Epub 2020 Jul 10. PMID 32871681
- [Background] de Aguiar Neto FS, Rosa JLG. Depression biomarkers using non-invasive EEG: A review. Neurosci Biobehav Rev. 2019 Oct;105:83-93. doi: 10.1016/j.neubiorev.2019.07.021. Epub 2019 Aug 7. PMID 31400570
- [Background] Brakowski J, Spinelli S, Dorig N, Bosch OG, Manoliu A, Holtforth MG, Seifritz E. Resting state brain network function in major depression - Depression symptomatology, antidepressant treatment effects, future research. J Psychiatr Res. 2017 Sep;92:147-159. doi: 10.1016/j.jpsychires.2017.04.007. Epub 2017 Apr 24. PMID 28458140
- [Background] Jesulola E, Sharpley CF, Agnew LL. The effects of gender and depression severity on the association between alpha asymmetry and depression across four brain regions. Behav Brain Res. 2017 Mar 15;321:232-239. doi: 10.1016/j.bbr.2016.12.035. Epub 2016 Dec 29. PMID 28042006
- [Background] Quraan MA, Protzner AB, Daskalakis ZJ, Giacobbe P, Tang CW, Kennedy SH, Lozano AM, McAndrews MP. EEG power asymmetry and functional connectivity as a marker of treatment effectiveness in DBS surgery for depression. Neuropsychopharmacology. 2014 Apr;39(5):1270-81. doi: 10.1038/npp.2013.330. Epub 2013 Nov 28. PMID 24285211
- [Background] Nusslock R, Shackman AJ, Harmon-Jones E, Alloy LB, Coan JA, Abramson LY. Cognitive vulnerability and frontal brain asymmetry: common predictors of first prospective depressive episode. J Abnorm Psychol. 2011 May;120(2):497-503. doi: 10.1037/a0022940. PMID 21381804
- [Derived] Wang Y, He WY, Zhan CAA, Pan SL, Wu W, Li FX, Zhang HF. Protocol for prognosticating PPD using EEG changes during labor pain by uterine contractions: a prospective cohort study in the first stage of labor. BMC Pregnancy Childbirth. 2025 Jan 22;25(1):49. doi: 10.1186/s12884-025-07167-1. PMID 39844134